CLINICAL TRIAL: NCT06170567
Title: The Effect of Crossword Puzzles on Nursing Students' Learning Concepts Related to Vital Signs: A Randomized Controlled Study
Brief Title: The Effect of Puzzles on Concept Learning in Nursing Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bilecik Seyh Edebali Universitesi (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Aysun Acun 2
Record Dates: First submitted 2023-12-04; First posted 2023-12-14 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2023-12

CONDITIONS: Students, Nursing; Education, Nursing
Keywords: Nursing students; puzzles; teaching

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Students' course success (Experimental): The effect of puzzles on students' course success
  Interventions: Other: The effect of puzzles on students' course success
- Student scores (Experimental): The effect of puzzles on students' course success
  Interventions: Other: The effect of puzzles on students' course success

INTERVENTIONS:
Other: The effect of puzzles on students' course success — The effect of puzzles on students' course success

SUMMARY:
Vital signs are concepts that first-year nursing students learn for the first time. Students are afraid of making mistakes in the concepts they are trying to learn for the first time. Learning and measuring vital signs are among the duties, powers and responsibilities of the nurse. Therefore, it is important for students to understand and learn correctly. At this point, puzzles are of great importance as they make learning easier and entertaining. The entertaining education of puzzles reduces students' fear of mistakes regarding concepts. This study aimed to investigate the effect of puzzles on nursing students' learning concepts related to vital signs.

DETAILED DESCRIPTION:
Puzzles, which are among the active learning tools, are frequently preferred today because they make learning fun, are economical, improve problem-solving skills and offer understandable learning. Puzzles increase students' motivation and self-confidence by turning complex concepts into a hobby. In the literature, studies investigating the learning situation with puzzles have examined undergraduate students in different sciences. Even though there are different disciplines, undergraduate students' efforts to search for the right answer, their self-confidence in finding the right answer, and their involvement in the active learning process rather than passive memorization reveal the increase in their knowledge levels. It has been observed that the teaching method with puzzles not only facilitates learning, but also guides students to better recognize their knowledge gaps and weaknesses. Considering nursing education, it is obvious that teaching concepts encountered for the first time with puzzles by providing an active environment in the classroom will increase students' motivation and knowledge level. Despite research conducted with different disciplines in the literature, there are few studies examining the effect of puzzles on the level of learning concepts related to the nursing profession. In this research, the concepts of vital signs, which have an important place in both the student life and professional life of first-year nursing students, will be discussed. An active and fun environment will be provided to students with puzzles on the subjects of respiration, pulse and blood pressure, where students have difficulty in learning the conceptual structure. In this context, it is predicted that the education provided with puzzles will contribute positively to the knowledge level of the students.

A pre-test will be given to all groups before the theoretical lesson on vital signs. Afterwards, the students in the experimental group will apply puzzles for two weeks (12-27/11/2023). Afterwards, final tests will be performed. The work will continue until 10/12/2023.

Control group students will be educated only during the normal course. The research will be conducted with first-year students of Bilecik Şeyh Edebali University Nursing Department.

ELIGIBILITY:
Inclusion Criteria:

* Being a first year nursing student a
* Taking a course on vital signs for the first time
* Volunteering to participate in research.

Exclusion Criteria:

*Not volunteering to participate in the research

Min Age: 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2023-12-20 (Actual); Study Completion 2024-01-10 (Actual)

PRIMARY OUTCOMES:
Student scores | 5 weeks
  Students' knowledge test successes will be seen.

CONTACTS AND LOCATIONS:
Locations (1):
- Bilecik Şeyh Edebali University, Bilecik, Turkey (Türkiye)